CLINICAL TRIAL: NCT01567657
Title: Phase II Study of Comparison of Two Sedation Regimen for Transesophageal Echocardiography in Point of View of Blood Pressure Response, Safety and Patient Comfort
Brief Title: Safety Study of Two Regimen for Sedation for Transesophageal Echocardiography
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kantonsspital Münsterlingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: TEE 2012
Record Dates: First submitted 2012-01-04; First posted 2012-03-30 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Hypotension
Keywords: Sedation in TEE; Blood pressure drop during TEE; Safety of sedation in TEE
MeSH Terms: conditions — Hypotension | interventions — Midazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pethidin plus midazolam (Active Comparator): Initial dose of 25 mg Pethidin iv. plus 1-2 mg Midazolam iv. Additional Bolus of Midazolam (1 mg wise iv.) if needed, until a maximal dose of 7 mg Midazolam iv.
  Interventions: Drug: Propofol
- Propofol (Active Comparator): Initial dose of Propofol of 50-60 mg iv. for patients 50 years or younger. Initial dose of Propofol of 30-40 mg iv. for patients over 50 years. If needed additional Bolus of 20-30 mg Propofol iv. as usual until sedation is achieved.
  Interventions: Drug: pethidin hydrochlorid, midazolam

INTERVENTIONS:
Drug: pethidin hydrochlorid, midazolam — Pethidin hydrochlorid: 25 mg iv. at the beginning of the examination Midazolam: 1-2 mg iv. at the beginning of the examination. Repetitive given in a dosis of 1 mg iv. until a total amount of 7 mg iv.
  Other Names: Pethidin hydrochlorid = Meperidine (USA); Midazolam = Dormicum
  Arms: Propofol
Drug: Propofol — 50 years and over: initial dose of 50-60 mg Propofol iv. Followed by bolus of 20-30 mg iv. until sedation is achieved.
  < 50 years: initial dose 30-40 mg Propofol iv. Followed by bolus of 10-20 mg until sedation is achieved.
  Other Names: Propofol = Propofolum = Diprivan = Disoprivan
  Arms: Pethidin plus midazolam

SUMMARY:
The purpose of this study is to determine whether sedation with a combination of pethidin hydrochlorid plus midazolam intravenously (i.v.) is superior to propofol i.v. alone in relation to blood pressure drops during an transesophageal echocardiographic examination (TEE).

DETAILED DESCRIPTION:
Randomisation is done immediately after information of the patient and obtaining of the informed consent. The average time for a TEE study is about 30 minutes. Data collection occurs during this time frame. ECG monitoring and data collection (blood pressure, heart rate, SO2) for the study protocol starts 6 minutes before the application of the sedation. At -6, -4, -2 minutes before the application of the sedation, baseline data are collected. The average systolic blood pressure of these three measures is taken as the reference blood pressure. This is the reference value to calculate the blood pressure drop during the examination. Blood pressure, pulse oxymetry, heart rate are taken every 2 minutes until the examination (TEE) is finished. The questionnaire (for second end points) is filled out by the patient within two hours after the examination. The patient will be followed for the duration of about one hour after the examination, if he is from the outpatient clinic. Patients from the hospital (inpatients) will be followed routinely in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* all patients scheduled for TEE in our department who have signed the informed consent except those younger than 18 years and patients with a second or third etc. TEE

Exclusion Criteria:

* < 18 years
* intensive care patients
* emergency department patients
* breast feeding women
* pregnant women
* patients with an allergy to Propofol or its ingredient soy oil, Pethidin or Midazolam

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with a blood pressure drop of more than 30 mmHg and below 100 mmHg systolic | During examination (TEE), expected to be ca. 30 minutes

SECONDARY OUTCOMES:
Number of patients with adverse events | At time of transfer to the ward, expected to be after ca. 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Fritz Widmer, Dr. med., Study Director — Departement of Cardiology, Kantonsspital Münsterlingen
Locations (1):
- Kantonsspital Münsterlingen, Münsterlingen, Thurgau, Switzerland